CLINICAL TRIAL: NCT01943435
Title: A Comparison of Non-Surgical Treatment Methods for Patients With Lumbar Spinal Stenosis
Brief Title: Study Comparing 3 Different Treatments for Arthritis of the Lower Back (Lumbar Spinal Stenosis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Schneider, DC, PhD (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Michael Schneider, DC, PhD, Assistant Professor, Department of Physical Therapy, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO12120422; 587 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2013-09-08; First posted 2013-09-17 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Spinal Stenosis; Spinal manipulation; Exercise; Epidural injection
MeSH Terms: conditions — Spinal Stenosis; Motor Activity | interventions — Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen; Celecoxib; Diclofenac; Misoprostol; Acetaminophen; Tramadol; Gabapentin; Nortriptyline; Duloxetine Hydrochloride; Sertraline; Trazodone; Mirtazapine; Papaverine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medical Care (Active Comparator): Non-steroidal anti-inflammatory drugs (NSAIDs); adjunctive analgesics; adjunctive anti-depressants. Participants assigned to this group will see a board certified physical medicine and rehabilitation physician for a history and examination, after which a determination will be made about a course of treatment that involve medications that are individualized to the needs of each patient.
  * NSAIDs: ibuprofen, celecoxib, or diclofenac/misoprostol
  * Adjunctive analgesics: acetaminophen, tramadol, or gabapentin
  * Adjunctive antidepressant agents: nortriptyline, duloxetine, sertraline, trazodone, or mirtazapine
  Lumbar epidural injection: these will be prescribed by the physician if warranted due to severity of symptoms or lack of adequate response to oral medications.
  Interventions: Drug: NSAIDs; adjunctive analgesics; adjunctive anti-depressants; Procedure: Lumbar epidural injection
- Group Exercise (Active Comparator): Group Exercise: community setting. This arm will involve attendance at community based group exercise classes that are taught by senior physical fitness instructors. These classes are designed specifically for older adults. Exercise frequency will be 2 times per week, for a total of 12 visits over the 6-week research period. These exercise classes will be attended at local community senior centers which cater to the needs of older adults. The subjects can self-select which particular exercise class they prefer to attend, based upon their level of fitness and physical function.
  Interventions: Other: Group Exercise: community setting
- Manual therapy and exercise (Active Comparator): This group of subjects will be treated with a combination of manual therapy and rehabilitative exercise procedures that are commonly used in the physical therapy and chiropractic professions. Subjects will be treated at a frequency of 2 times per week, for a total of 12 visits over the 6-week research period. Treatments will be provided by licensed physical therapists and chiropractors using a combination of Joint Mobilizations (spine, sacroiliac, hip), muscle stretching and strengthening exercises.
  Individualized exercises: clinical setting. These exercises will be tailored to the individual needs of each research participant by the treating physical therapist or chiropractor.
  Interventions: Other: Joint Mobilizations (spine, sacroiliac, hip); Other: Individualized exercises: clinical setting

INTERVENTIONS:
Drug: NSAIDs; adjunctive analgesics; adjunctive anti-depressants — Physician will administer these medications based upon the individual needs of each patient.
  Other Names: ibuprofen; celecoxib; diclofenac; misoprostol; acetaminophen; tramadol; gabapentin; nortriptyline; duloxetine; sertraline; trazodone; mirtazapine
  Arms: Medical Care
Procedure: Lumbar epidural injection — The attending physician may refer subjects for epidural injections at a pain clinic that is affiliated with the University of Pittsburgh Medical Center. All epidural injections will be provided by licensed physicians who are board certified in physical medicine and rehabilitation or anesthesiology.
  Arms: Medical Care
Other: Joint Mobilizations (spine, sacroiliac, hip) — These joint mobilizations will be applied manually to the lumbar facet joints, sacroiliac joints, and/or hip joints by licensed physical therapists and chiropractors.
  Arms: Manual therapy and exercise
Other: Individualized exercises: clinical setting — The treating physical therapist or chiropractor will work with each subject to develop a set of individualized exercises in the clinic setting. The goal is to have the subjects continue these exercises at home.
  Arms: Manual therapy and exercise
Other: Group Exercise: community setting — The group exercise will take place at community centers that provide exercise classes for older adult. The exercises are taught by certified fitness instructors in a group setting at these community centers.
  Arms: Group Exercise

SUMMARY:
BACKGROUND: Lumbar spinal stenosis - known by patients as "arthritis of the spine" - is a condition that is very common; found in about 30% of older adults. It is the most common reason for people over the age of 65 to have back surgery. Some patients with stenosis do not need back surgery and can be treated with other methods, such as physical therapy, chiropractic, exercise, and medication. But we just don't have enough good research to tell us which treatment works best for which patient and under which circumstances. This research study hopes to provide more information about the effectiveness of the various non-surgical choices for managing stenosis.

OBJECTIVES: This study will directly compare the effectiveness of three common non-surgical treatment approaches for stenosis:

1. Medical care that involves prescription medications and/or spinal injections (epidurals)
2. Group exercise in supervised classes given in a community center setting
3. Hands-on (manual) therapy and rehabilitative exercises given in a clinic setting by physical therapists and chiropractors

METHODS: This research study will involve 259 adults who are at least 60 years old and have been diagnosed with lumbar spinal stenosis. The research volunteers will be divided into three groups, each group receiving one of the 3 types of treatments listed above under "Objectives". The determination of which type of treatment each person receives will be determined by chance, using a computerized version of flipping a coin. This is a process known as randomization, which scientists think reduces the bias in research studies. A series of tests and questionnaires will be given to the patients before and after they get treatment and comparisons will be made to see how much improvement they made with each of the types of treatments. Finally, the researchers will compare the differences between the 3 treatment groups to see if certain types of treatment produced better results than others, and if there were any examination findings that could be used to predict which type of patient would do better with which type of treatment.

DETAILED DESCRIPTION:
BACKGROUND: Lumbar spinal stenosis (LSS) is a condition that is highly prevalent in the senior citizen population. LSS is the most frequent indication for spinal surgery in patients over the age of 65 years. The fastest growth in lumbar surgery in the U.S. this past decade has occurred in older adults with LSS and the rate of complex fusion procedures has increased 15-fold. These surgical procedures are associated with significant health care costs, risks, complications, and re-hospitalization rates. Yet, evidence is lacking for the effectiveness of the various non-surgical treatments offered to patients with LSS. This knowledge gap has greatly hindered the development of clinical practice guidelines relevant to the non-surgical treatment approaches for LSS.

OBJECTIVES: This study will perform a comparison of three common approaches to the non-surgical management and treatment of patients with LSS. The specific research questions associated with this study are: (1) How do group exercise and manual therapy with rehabilitative exercise compare with medical care? (2) How do group exercise and manual therapy with rehabilitative exercise compare with each other? (3) Are there any baseline predictors associated with clinical improvement in any of these non-surgical treatment approaches? The long term objective of this study is to produce research evidence relevant to community stakeholders and to inform better decision making about non-surgical treatment options available to LSS patients.

METHODS: This will be a comparative effectiveness study utilizing the research design of a randomized controlled clinical trial (RCT). It will be a 3-group RCT that allows for pragmatic treatment approaches in each of the three study arms. The study sample will consist of 259 older adults (>60 years) who have symptoms consistent with a diagnosis of LSS, which will be confirmed by clinical examination and diagnostic imaging. Eligible subjects will be randomized into one of three pragmatic treatment approaches: 1) medical care; 2) group exercise; or 3) manual therapy with rehabilitative exercise.

All subjects will be treated for a 6-week course of care. Primary outcome measures are two validated research measurement tools; the Swiss Spinal Stenosis Questionnaire (self-reported pain/function) and the Self Paced Walking Test (performance-based measure). We will also employ a novel secondary outcome measure; the Sense Wear Armband which provides a real-time measure of physical activity during normal daily living.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 60 years
* Can read/write English and understand directions
* Diagnosis of lumbar spinal stenosis confirmed by CT or MRI scan
* Has limitation of standing and/or walking tolerance
* Willing to attend treatments 2 times per week for 6 weeks
* Ability to walk at least 50 feet without the need for a cane or walker

Exclusion Criteria:

* History of metastatic cancer
* Advised by a physician not to exercise
* History of lumbar surgery for spinal stenosis or previous lumbar fusion
* Presence of severe peripheral artery disease in legs
* Severe hypertension: Systolic > 200 mm/hg or Diastolic > 110 mm/hg
* Ankle brachial index < 0.8
* Neurologic or neurodegenerative disease other than stenosis that severly impairs the ability to walk
* Presence of cauda equina symptoms (saddle paresthesia, progressive loss of bladder/bowel function, etc)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Schneider, PhD, DC, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Center for Integrative Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other researchers at the discretion and approval of the PI.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Schneider M, Ammendolia C, Murphy D, Glick R, Piva S, Hile E, Tudorascu D, Morton SC. Comparison of non-surgical treatment methods for patients with lumbar spinal stenosis: protocol for a randomized controlled trial. Chiropr Man Therap. 2014 May 10;22:19. doi: 10.1186/2045-709X-22-19. eCollection 2014. PMID 24872875
- [Derived] Roseen EJ, Smith CN, Rahim A, Deal C, Fischer R, Morone NE, Flack A, Penza C, Suri P, Dougherty PE, Weiner DK, Schneider MJ. Which lumbar spinal stenosis patients will improve with nonsurgical treatment? A secondary analysis of a randomized controlled trial. Chiropr Man Therap. 2025 Dec 9;33(1):57. doi: 10.1186/s12998-025-00620-0. PMID 41366694
- [Derived] Schneider MJ, Ammendolia C, Murphy DR, Glick RM, Hile E, Tudorascu DL, Morton SC, Smith C, Patterson CG, Piva SR. Comparative Clinical Effectiveness of Nonsurgical Treatment Methods in Patients With Lumbar Spinal Stenosis: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jan 4;2(1):e186828. doi: 10.1001/jamanetworkopen.2018.6828. PMID 30646197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general population in the City of Pittsburgh from November 2013 through November 2015.
Pre-assignment Details: We consented and randomized a total of 259 subjects. However, 19 of those randomized subjects who never received any treatment...i.e. they dropped out after randomization but before their first scheduled treatment. Therefore, we a total of 240 subjects who were actually enrolled and received at least one treatment.
Groups:
- Medical Care: Participants assigned to this group will see a board certified physical medicine and rehabilitation physician for a history and examination, after which a determination will be made about a course of treatment that involve medications that are individualized to the needs of each patient. These include any of the following:
  NSAIDs, Adjunctive analgesics, antidepressants,
  Lumbar epidural injection: prescribed by the physician if warranted due to severity of symptoms or lack of adequate response to oral medications. Shared decision making with patient.
- Manual Therapy and Exercise: This group of subjects will be treated with a combination of manual therapy and rehabilitative exercise procedures that are commonly used by physical therapists and chiropractors. Subjects will be treated at a frequency of 2 times per week, for a total of 12 visits over the 6-week research period. Treatments provided by licensed physical therapists and chiropractors include:
  Manual Therapy: Joint mobilizations of the lumbar spine, sacroiliac, and/or hip joints, as well as muscle stretching and neural mobilizations
  Rehabilitative exercises: exercises will be tailored to the individual needs of each research participant by the treating physical therapist or chiropractor.
Period: Baseline Eligibility and Randomization
Arm/Group | Medical Care | Group Exercise | Manual Therapy and Exercise
Started | 88 | 84 | 87
Completed | 84 | 72 | 84
Not Completed | 4 | 12 | 3
Not completed — Withdrawal by Subject | 4 | 12 | 3
Period: Intervention Period
Arm/Group | Medical Care | Group Exercise | Manual Therapy and Exercise
Started | 84 | 72 | 84
Completed | 81 | 69 | 80
Not Completed | 3 | 3 | 4
Not completed — Withdrawal by Subject | 3 | 3 | 4
Period: 2 Month Follow up
Arm/Group | Medical Care | Group Exercise | Manual Therapy and Exercise
Started | 81 | 69 | 80
Completed | 79 | 66 | 80
Not Completed | 2 | 3 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0
Period: 6 Month Follow up
Arm/Group | Medical Care | Group Exercise | Manual Therapy and Exercise
Started | 79 | 66 | 80
Completed | 67 | 59 | 65
Not Completed | 12 | 7 | 15
Not completed — Lost to Follow-up | 12 | 7 | 15

BASELINE CHARACTERISTICS:
Groups:
- Usual Medical Care: Participants assigned to this group will see a board certified physical medicine and rehabilitation physician for a history and examination, after which a determination will be made about a course of treatment that involve medications that are individualized to the needs of each patient. These include any of the following: NSAIDs, Adjunctive analgesics, antidepressants.
  Lumbar epidural injection: prescribed by the physician if warranted due to severity of symptoms or lack of adequate response to oral medications. Shared decision making with patient.
  Lumbar epidural injection: these will be prescribed by the physician if warranted due to severity of symptoms or lack of adequate response to oral medications.
  NSAIDs; adjunctive analgesics; adjunctive anti-depressants: Physician will administer these medications based upon the individual needs of each patient.
  Lumbar epidural injection: The attending physician may refer s
- Total: Total of all reporting groups
Arm/Group | Usual Medical Care | Group Exercise | Manual Therapy and Exercise | Total
Number analyzed (Participants) | 88 | 84 | 87 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (7.4) | 72.9 (8.1) | 72.1 (8.1) | 72.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 39 | 52 | 137
  Male | 42 | 45 | 35 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 88 | 84 | 87 | 259
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 19 | 18 | 19 | 56
  White | 68 | 66 | 67 | 201
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 88 | 84 | 87 | 259
Swiss Spinal Stenosis Total Score [Mean (Standard Deviation); unit: units on a scale] — The SSS is a patient self-reported measure of pain and function related to spinal stenosis. The total score range is 12-55 with increasing values representing worsening disability.
  units on a scale | 31.4 (5.8) | 31.6 (6.0) | 31.7 (6.1) | 31.5 (6.0)
Self Paced Walk Test Total Distance [Mean (Standard Deviation); unit: meters] | 482.2 (529.1) | 433.4 (421.2) | 449.2 (485.2) | 455.3 (480.0)

OUTCOME MEASURES:

1. Primary Outcome: Swiss Spinal Stenosis (SSS) Questionnaire Score
Description: Our primary aim included a primary outcome measure of self-reported pain/function, which was the change in SSS total score between baseline and 8 weeks. The Swiss Spinal Stenosis Questionnaire (SSS) is a validated 12-item condition-specific instrument for patients with lumbar spinal stenosis. It provides a patient self-report measure of pain and physical function. Higher scores represent worse symptoms and less physical function. The 12-item SSS total score range is 12-55. For our analysis, we compared the change in the 12-item Total score from baseline to 8 weeks.
Time Frame: Primary End-Point was 8 weeks ( 2 weeks after completion of 6-week intervention).
Population: Analysis performed on all randomized participants and linear mixed models were used to account for missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Manual Therapy and Exercise: This group of subjects will be treated with a combination of manual therapy and rehabilitative exercise procedures that are commonly used by physical therapists and chiropractors. Subjects will be treated at a frequency of 2 times per week, for a total of 12 visits over the 6-week research period. Treatments provided by licensed physical therapists and chiropractors include:
  Manual Therapy: Joint mobilizations of the lumbar spine, sacroiliac, and/or hip joints, as well as muscle stretching and neural mobilizations.
  Rehabilitative exercises: exercises will be tailored to the individual needs of each research participant by the treating physical therapist or chiropractor.
Arm/Group | Medical Care | Group Exercise | Manual Therapy and Exercise
Number analyzed (Participants) | 88 | 84 | 87
units on a scale | -2.0 (5.5) | -1.7 (5.2) | -4.1 (5.9)
Statistical Analysis 1: Comparison: Medical Care vs Group Exercise; The primary analysis was a between-groups comparison of means using linear mixed models with SSS total score as the dependent variable, while adjusting for randomization stratification factors; Test type: Superiority — For this superiority study, sample size estimation was based upon hypothesized changes in our primary outcome measure, the Swiss Spinal Stenosis (SSS) questionnaire. We calculated that a total sample size of 180 subjects (n=60 per group) would give us 80% power to detect a difference as small as 3.6 points on the Swiss Spinal Stenosis questionnaire score. Sample size was increased at the request of the funding agency without any interim analysis performed; p = 0.73, Regression, Linear; Linear mixed models were adjusted for randomization stratification factors; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.5 to 2.2]
Statistical Analysis 2: Comparison: Medical Care vs Manual Therapy and Exercise; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.02, Regression, Linear; Linear mixed models were adjusted for randomization stratification factors; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-3.9 to -0.3]
Statistical Analysis 3: Comparison: Group Exercise vs Manual Therapy and Exercise; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.01, Regression, Linear; Linear mixed models were adjusted for randomization stratification factors; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [0.6 to 4.3]

2. Secondary Outcome: Self Paced Walking Test (SPWT)
Description: Our primary aim also included a performance-based outcome measure, which was the distance walked during the SPWT. The analysis was a comparison of between-group changes in SPWT between baseline and 8 weeks. The Self-Paced Walking Test (SPWT) is a validated objective measure of a patient's walking capacity, which is performed on a level walking surface. The patient is instructed to walk at their own pace and to stop when the symptoms are troublesome enough that s/he needs to sit down to rest. The total time and total distance walked are measured by the research assistant. Our unit of measure was the total distance walked, expressed in meters.
Time Frame: Primary end-point was 8 weeks ( 2 weeks after 6 week intervention is completed).
Population: Analysis performed on all randomized participants and linear mixed models were used to account for missing data.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Medical Care | Group Exercise | Manual Therapy and Exercise
Number analyzed (Participants) | 88 | 84 | 87
meters | 130.5 (478.7) | 219.2 (413.0) | 267.8 (507.8)
Statistical Analysis 1: Comparison: Medical Care vs Group Exercise; This analysis consisted of a between-groups comparison of means using linear mixed models with SPWT as the dependent variable, while adjusting for randomization stratification factors; Test type: Superiority; p = 0.29, Regression, Linear; Linear mixed models were adjusted for randomization stratification factors; Mean Difference (Final Values) = 87.0, 95% CI 2-sided [-75.2 to 249.2]
Statistical Analysis 2: Comparison: Medical Care vs Manual Therapy and Exercise; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.10, Regression, Linear; Linear mixed models were adjusted for randomization stratification factors; Mean Difference (Final Values) = 129.7, 95% CI 2-sided [-27.2 to 286.6]
Statistical Analysis 3: Comparison: Group Exercise vs Manual Therapy and Exercise; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.61, Regression, Linear; Linear mixed models were adjusted for randomization stratification factors; Mean Difference (Final Values) = -42.7, 95% CI 2-sided [-205.4 to 120.0]

3. Other Pre Specified Outcome: Sense Wear Armband
Description: Our secondary aim was to measure the change in physical activity between baseline and 8 weeks using the Sense Wear armband (SWA). The outcome measure was the average number of minutes spent daily performing physical activities >1.5 metabolic equivalents (METs).The SWA is a small device that collects information from multiple sensors: a triaxial accelerometer, heat flux, skin temperature, and galvanic signal. The information is integrated and processed by software using proprietary algorithms utilizing subjects' demographic characteristics (gender, age, height, and weight) to provide minute-by-minute estimates of physical activity. The SWA has shown good reliability and validity. The research participants in our study will wear the SWA for a week before and after they complete the treatment interventions.
Time Frame: Primary End-Point was 8 weeks ( 2 weeks after completion of 6-week intervention).
Population: Analysis performed on all randomized participants and linear mixed models were used to account for missing data.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Medical Care | Group Exercise | Manual Therapy and Exercise
Number analyzed (Participants) | 88 | 84 | 87
minutes per day | -23.1 (85.3) | 4.3 (64.8) | -6.0 (76.0)
Statistical Analysis 1: Comparison: Medical Care vs Group Exercise; This secondary analysis consisted of a between-groups comparison of means using linear regression with physical activity as the dependent variable (average number of minutes spent daily in activities >1.5 METs), while adjusting for randomization stratification factors; Test type: Superiority; p = 0.03, Regression, Linear; Linear mixed models were adjusted for randomization stratification factors; Mean Difference (Final Values) = 30.5, 95% CI 2-sided [3.1 to 57.9]
Statistical Analysis 2: Comparison: Medical Care vs Manual Therapy and Exercise; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.16, Regression, Linear; Linear mixed models were adjusted for randomization stratification factors; Mean Difference (Final Values) = 18.7, 95% CI 2-sided [-7.6 to 45.0]
Statistical Analysis 3: Comparison: Group Exercise vs Manual Therapy and Exercise; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.40, Regression, Linear; Linear mixed models were adjusted for randomization stratification factors; Mean Difference (Final Values) = 11.8, 95% CI 2-sided [-15.6 to 39.1]

ADVERSE EVENTS:
Time Frame: Assessed from beginning of treatment up to 2 month follow up assessment.
Groups:
- Medical Care: Participants assigned to this group will see a board certified physical medicine and rehabilitation physician for a history and examination, after which a determination will be made about a course of treatment that involve medications that are individualized to the needs of each patient. These include any of the following: NSAIDs, Adjunctive analgesics, antidepressants.
  Lumbar epidural injection: prescribed by the physician if warranted due to severity of symptoms or lack of adequate response to oral medications. Shared decision making with patient.
Arm/Group | Medical Care | Group Exercise | Manual Therapy and Exercise
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/72 | 0/84
Other Adverse Events (participants affected / at risk) | 18/84 | 25/72 | 54/84
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Care (N=84) | Group Exercise (N=72) | Manual Therapy and Exercise (N=84)
Gastrointestinal Symptoms (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0)
Drowsiness (General disorders) | 5 (5) | 0 (0) | 0 (0)
Dry Mouth (General disorders) | 4 (4) | 0 (0) | 0 (0)
Joint soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (10) | 40 (93)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 5 (5) | 22 (26) | 44 (115)

LIMITATIONS AND CAVEATS:
We realize in retrospect that our original choice of the term "usual medical care" may have been confusing, because there is great variation in the medical management of patients with stenosis. We suggest that "medical care" is a better term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes